CLINICAL TRIAL: NCT06978075
Title: Research on the Application of Artificial Intelligence (AI) Assisted Chest Wall Tumor Resection Combined With Personalized 3D Preformed Chest Wall Defection Reconstruction System in Chest Wall Tumor Surgery
Brief Title: Artificial Intelligence Combined With 3D-Preformed Chest Wall Defection Reconstruction System in Chest Wall Tumor Surgery
Acronym: AICW3DPCWDRS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wu Weiming (Other)
Responsible Party: Sponsor-Investigator, Wu Weiming, Shanghai Jiao Tong University Affiliated Sixth People's Hospital of medicine, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Organization: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240910
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Chest Wall Tumor; Reconstruction Surgery
Keywords: chest wall tumor resection and reconstrucion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chest wall tumor (Experimental)
  Interventions: Device: Chest wall tumor resection by the artificial intelgent assistent

INTERVENTIONS:
Device: Chest wall tumor resection by the artificial intelgent assistent — we plan to carry out of the research on the application of artificial intelligence (AI) assisted chest wall tumor research combined with a personalized 3D preformed chest wall defect reconstruction system in chest wall tumor surgery. Data will be imported into a computer to draw a 3D model of the tumor and construct an ideal resection range to ensuring sufficient surgical margins while avoiding damage to important nerve and vascular tissues in the chest. Preformed titanium plates will be prepared based on the calculated resection range and the titanium plates will be detachable assembly components through screws, which can be adjusted at any time according to the surgical situation.

SUMMARY:
Chest wall tumors should be completely resection as much as possible while malignant chest wall tumors should be extensively resection. If not completely resection, it will recur in the short time and affect the patient's survival. At present, the surgical resection range mainly relies on preoperative imaging examination and the experience of the surgeon. It lacks precise guidance. This can easily lead to incomplete resection. In addition, the reconstruction materials required for reconstruct the excised chest wall defection are often generated in a standardized manner, lacking intraoperative adjustability. To address this clinical issue, we plan to carry out the research on the application of artificial Intelligence (AI) assisted chest wall tumor resection combined with personalized 3D preformed chest wall defection reconstruction system in chest wall tumor surgery.

DETAILED DESCRIPTION:
Chest wall tumors should be completely removed as much as possible while malignant tumors should be extensively resection. Due to the lack of sensitivity of the vast majority of chest wall malignant tumors to current chemotherapy drugs, radiotherapy techniques, and even targeted drugs. If not completely resected, the tumor may recur in the short time and catastrophic consequences may occur. At present, the surgical resection range mainly relies on traditional imaging examinations before surgery and the clinical experience of the surgeon. It lacks precise instrument or equipment guidance. This can easily lead to incomplete surgical resection range. In addition, for the reconstruction materials required to reconstruct the chest wall defection after resection, they are often produced in a standardized manner and need to be adjusted according to the surgical situation. Even with 3D printed titanium alloy materials currently available, there is a possibility that they may not be usable once the lesion area exceeds preoperative assessment. To address this clinical issue, we plan to carry out of the research on the application of artificial intelligence (AI) assisted chest wall tumor research combined with a personalized 3D preformed chest wall defect reconstruction system in chest wall tumor surgery. Data will be imported into a computer to draw a 3D model of the tumor and construct an ideal resection range to ensuring sufficient surgical margins while avoiding damage to important nerve and vascular tissues in the chest. Preformed titanium plates will be prepared based on the calculated resection range and the titanium plates will be detachable assembly components through screws, which can be adjusted at any time according to the surgical situation.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old, male or female not limited
2. Anesthesia ASA score I-II
3. Malignant tumor of soft tissue in the chest
4. Malignant tumors of ribs, rib cartilage, and sternum
5. Tumors with uncertain or unknown properties of ribs, rib cartilage, and sternum
6. Giant benign tumors of ribs, rib cartilage, and sternum
7. The preoperative examination results indicate that the tumor has not undergone distant metastasis
8. Willing to participate in the research and sign the informed consent form

Exclusion Criteria:

1. Patients with distant metastasis detected during preoperative examination
2. Inoperable tumor
3. During the examination, it was discovered that the patient had another type of malignant tumor present
4. ECOG 4
5. Suffering from active or chronic fungal/bacterial/viral infections
6. History of allergy to anesthesia related drugs
7. Heart and lung dysfunction, liver and kidney dysfunction, inability to tolerate surgery
8. Patients with mental disorders who are unable to cooperate with treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
the tumor status of surgical margin | 3 year
  Visible tumor residue with naked eye, tumor cells visible under microscope, no tumor cells observed under microscope

SECONDARY OUTCOMES:
Stability after chest wall reconstruction | 3 year
  3D pre formed titanium plates are used for chest wall defect reconstruction. Based on the size and shape of the defect during surgery, suitable titanium plates are selected and fixed with nooses for chest wall defect reconstruction surgery.

IPD SHARING:
Plan to Share IPD: No